CLINICAL TRIAL: NCT00006498
Title: Chronic Life Stress and Incident Asthma in Adult Women
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Other Study IDs: 939; R01HL064108 (NIH)
Record Dates: First submitted 2000-11-16; First posted 2000-11-17 (Estimated); Last update posted 2016-03-16 (Estimated); Status verified 2006-01

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases

SUMMARY:
To prospectively examine the association between a specific chronic life stressor (i.e., intimate violence exposure) and adult asthma in women.

DETAILED DESCRIPTION:
BACKGROUND:

Etiologies of the rising prevalence and morbidity of asthma are not well understood. Knowledge gaps are particularly significant with respect to adult-onset asthma. The role of stress in the expression of asthma is largely unexplored in large-scale, prospective, epidemiologic studies and such investigation has been identified as a priority by a recent NHLBI expert panel.

DESIGN NARRATIVE:

The study prospectively examines the association between a specific chronic life stressor (i.e., intimate violence exposure) and adult asthma in women participating in the Nurses' Health Study II cohort. Emerging epidemiologic data suggest that exposure to intimate violence is a pervasive chronic life stressor associated with adverse impact on womens' psychological and physical health. Traumatic stress such as that related to intimate violence exposure has been associated with neuroendocrine changes known to cause alterations in neuroendocrine and immune functions important to the pathophysiology of inflammatory diseases including asthma. The investigators are testing the hypothesis that women exposed to high-level chronic stress (violence) will be at greater risk for asthma development than women with low-level stress (violence) exposure. The influence of chronic stress on neuroendocrine and immune function as reflected in morning cortisol expression, for the former, and cytokine profiles and IgE production (T-helper cell polarization), for the latter, will also be examined in a nested case control fashion among these women.

The study completion date listed in this record was obtained from the "End Date" entered in the Protocol Registration and Results System (PRS) record.

ELIGIBILITY:
No eligibility criteria

Max Age: 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2000-09; Study Completion 2005-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rosalind Wright — Brigham and Women's Hospital